CLINICAL TRIAL: NCT02431429
Title: Spermiogram Assessment in Bolivian Patients Taking Impavido® (Miltefosine) for Mucocutaneous Leishmaniasis
Status: Completed | Type: Observational
Sponsor: Knight Therapeutics (USA) Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MILT 2127-2
Record Dates: First submitted 2015-04-22; First posted 2015-05-01 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2018-03

CONDITIONS: Mucocutaneous Leishmaniasis
Keywords: leishmaniasis; miltefosine; spermiogram
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis | interventions — miltefosine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- miltefosine: miltefosine: target of 2.5 mg/kg/day for 28 days
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine

SUMMARY:
This study is a Phase 4, open-label, single group study in which at least 55 evaluable adult male patients undergoing miltefosine treatment for mucocutaneous leishmaniasis will provide semen samples for spermiogram analysis of sperm parameters.

DETAILED DESCRIPTION:
This study is a Phase 4, open-label, single group study in which at least 55 evaluable adult male patients undergoing miltefosine treatment for mucocutaneous leishmaniasis will provide semen samples for spermiogram analysis of sperm parameters. Potential subjects diagnosed with mucocutaneous leishmaniasis who are planning to undergo miltefosine treatment will be informed about the study and undergo the informed consent process. After obtaining informed consent, subjects will be screened over a 28-day period for eligibility by medical history including leishmaniasis diagnostics, physical examination, clinical laboratory measurements [chemistries: (ALT, total bilirubin, creatinine; hematology: WBC count, hemoglobin, platelet count; spermiogram: sperm concentration, total sperm count, semen volume, sperm motility, and sperm morphology; hormones: testosterone and FSH]; and medication use in the 28-day period before starting treatment. If eligible for the study, the subject will receive miltefosine for 28 days at a target dose of approximately 2.5 mg/kg/day. Screening and enrollment into the study will continue until at least 55 subjects complete the study and are considered evaluable (provide sperm samples per protocol and complete at least 25 of 28 days of miltefosine treatment). Chemistries and hematology will be repeated at study Days 14 (mid-treatment) and 28 (end of treatment). Two semen samples will be collected during screening (at least 48 hours apart), at the end of treatment (Days 25-and-28), at 3-months after completing treatment. If clinically significant changes spermiogram findings are observed at 3 months, one sample will be collected at 6 months. Adverse events (AEs) and concomitant medication use will be collected during treatment. Concomitant medication use will also be collected at the 3-month visit and in any subject coming back for the 6-month visit. A medical history will be taken at the 3-month and 6-month (if conducted) focusing on any changes to the urogenital system.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Be available to complete study procedures
3. Have a diagnosis of mucocutaneous leishmaniasis confirmed by microscopy of a stained smear of a lesion sample, by culture of a lesion sample, or by polymerase chain reaction (PCR) of a lesion sample or by Montenegro skin test and be planning to undergo treatment with miltefosine
4. Be male and 18-55 years of age
5. Have ALT, total bilirubin, and creatinine < 1.5 upper limit of normal (ULN)
6. Have values of ions that might affect ECG (magnesium, calcium, potassium, sodium) within normal laboratory limits (WNL)
7. Have WBC count, hemoglobin, and platelet count within 15% of normal laboratory limits (WNL)
8. Have no known history of male sexual dysfunction
9. Have not had a vasectomy and agree to not have a vasectomy for the duration of the study
10. Have testosterone WNL (> 300 ng/dL) and FSH WNL (1.5 - 2.4 mIU/mL)
11. Have screening semen parameters (mean of both tests) of:

    1. semen volume at least 1.5 mL
    2. total sperm count greater than 45 million
    3. sperm concentration greater than 30 million/mL
    4. sperm motility greater than 50% (total percentage progressively motile sperm)
    5. normal sperm morphology by strict criteria >10%

Exclusion Criteria:

1. Have presence of any psychological or physiological abnormalities that in the opinion of the Investigator would significantly impair sexual performance or ability to provide semen samples according to the protocol
2. Have evidence by history of psychotropic and central nervous system drugs (e.g., antidepressants, anti-epileptics), anti-hypertensives, calcium channel blockers, chemotherapy drugs, colchicine, therapeutic hormones, finasteride, sulfasalazine, use of nicotine containing products or urine toxicology test for marijuana (tetrahydrocannabinol) and cocaine.
3. Have history of surgical prostatectomy
4. Have positive serology for Chagas Disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: mucocutaneous leishmaniasis patients
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
number of patients with abnormal spermiogram | 4 weeks of therapy plus up to 3-6 months after therapy

SECONDARY OUTCOMES:
number of patients with abnormal values of testosterone/FSH | 4 weeks of theapy plus up to 3-6 months after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Soto, MD, Principal Investigator — Fundacion Nacional de Dermatologia
Locations (1):
- Funderama, Santa Cruz, Bolivia